CLINICAL TRIAL: NCT04660721
Title: A Phase I/II, Randomized, Prospective, Controlled, Multi-center, Open-label, Two-arm Study Evaluating the Safety and Preliminary Efficacy of sFilm-FS in Controlling Liver Bleeding During Elective Surgery
Brief Title: A Study Evaluating the Safety and Preliminary Efficacy of sFilm-FS in Controlling Parenchymal Bleeding During Elective Hepatic Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sealantium Medical Ltd. (Industry)
Collaborators: Sintesi Research Srl (Industry); Home Medics Consulting Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEM-01-17
Record Dates: First submitted 2020-11-12; First posted 2020-12-09 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Hemostasis; General Surgery
Keywords: Body fluid leakage; Liver; Parenchymal bleeding; Hepatic surgery; Fibrin sealant; Fibrin patch; Human Fibrinogen; Human Thrombin; Coagulation
MeSH Terms: conditions — Thrombosis | interventions — TachoSil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- sFilm-FS (Experimental)
  Interventions: Combination Product: sFilm-FS
- TACHOSIL® (Active Comparator)
  Interventions: Combination Product: TACHOSIL®

INTERVENTIONS:
Combination Product: sFilm-FS — sFilm-FS is a sterile bio-compatible bio-absorbable patch embedded with lyophilized powders of Human Fibrinogen, Human Thrombin and calcium chloride.
  Arms: sFilm-FS
Combination Product: TACHOSIL® — TACHOSIL® is a fibrin sealant patch composed of an equine collagen patch coated with Human Fibrinogen and Human Thrombin.
  Arms: TACHOSIL®

SUMMARY:
The Study investigates a new product, sFilm-FS, aimed to help controlling body fluid leakage in general surgery procedures, proposing its use as an adjunct to hemostasis and/or sealing.

DETAILED DESCRIPTION:
Many products have been developed as adjuncts to hemostasis in bleeding situations where traditional methods such as suture, clips or energy-based coagulation are ineffective or impractical.

Many products are not as effective in the presence of active and/or brisk bleeding since the lack of sufficient adhesion strength allows forceful bleeding to simply "float" the products away from the bleeding tissue, prior to the achievement of full hemostasis.

The Study investigates a new product, sFilm-FS, aimed to help the control of body fluid leakage in general surgery procedures, proposing its use as an adjunct to hemostasis and/or sealing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (males or females) aged ≥ 18 years old.
2. Patients requiring elective open hepatic surgery.
3. Hemoglobin ≥ 8.0 g/dL within 24 hours prior to surgical procedure.
4. Patients understanding the nature of the study and providing their informed consent prior to participation.
5. Patients willing to participate in the study and able to attend the visits and procedures foreseen by study protocol.

   Intra-operative inclusion criteria:
6. Patients with a target bleeding site (TBS) identified by the Investigator during hepatic surgery (intra-operative inclusion criteria).

Exclusion Criteria:

1. Patients having undergone a therapeutic surgical procedure within 30 days from the study enrolment.
2. Patients with a severe coagulopathy defined as INR > 2.0.
3. Patients with platelet count <50,000 x109 PLT/L at the screening.
4. Patients admitted to trauma surgery.
5. Transplant patients due to fulminant hepatic failure.
6. Patients with known or suspected allergy or hypersensitivity to blood products or to one of the components of sFilm-FS or the active-comparator.
7. Patients with anesthesia risk judged to be higher than ASA3 by the Investigator.
8. Patients with at least one of the following concomitant conditions: severe co-morbid conditions known to pose a high risk for surgery and adequate recovery (i.e., liver cirrhosis with Child-Pugh score B or C, cholestasis, heart diseases), immunodeficiency diseases, blood clotting disorders, any conditions known to effect wound healing (i.e., collagen vascular disease), known or current alcohol or drug abusers.
9. Patients suffering from claustrophobia.
10. Patients with implanted or embedded metal objects, prostheses, pacemaker, or fragments in the head or body that would present a risk during the MRI scanning procedure or have worked with ferrous metals either as a vocation or hobby or following trauma (i.e., sheet metal workers, welders, or machinists) in such a way that might have led to unknown, indwelling metal fragments that could cause injury if they moved in response to placement in the magnetic field.
11. Patients being treated with at least one of the following treatments: antibiotic therapy for active infection, fibrin sealants, systemic steroids, or immunosuppressive agents.
12. Patients who are participating or have participated in other clinical studies within the 30 days before the study enrolment.
13. Female patients who are pregnant or breast-feeding or who wish to become pregnant during the period of the clinical study and for three months later.
14. Female patients of childbearing age (less than 24 months after the last menstrual cycle) who do not use adequate contraception.

    Intra-operative exclusion criteria:
15. Patients identified with a TBS with major arterial bleeding requiring suture or mechanical ligation.
16. Patients identified by the Investigator to have intra-operative bleeding from large defects in large arteries or veins, requiring repair.
17. Patients identified by the Investigator to have intra-operative findings that may preclude conduct of study procedure.
18. Patients having an active local infection in the anatomic surgical area.
19. Patients with occurrence of major intra-operative complications that require resuscitation or deviation from the planned surgical procedure.
20. Patients with bleeding site in or near to foramina in bone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orgad Laub, Professor, Study Director — Sealantium Medical Ltd.
Locations (4):
- Washington University in St. Louis, School of Medicine, Department of Surgery, St Louis, Missouri, United States
- Austria (2):
  - Ordensklinikum Linz GmbH Barmherzige Schwestern, Linz
  - Medical University of Vienna, Department of Surgery Hepatobiliary Unit, Vienna
- University Medical Center of Ljubljana, Division of Surgery, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spotnitz WD. Fibrin sealant: past, present, and future: a brief review. World J Surg. 2010 Apr;34(4):632-4. doi: 10.1007/s00268-009-0252-7. PMID 19820991
- [Background] Vonlanthen R, Slankamenac K, Breitenstein S, Puhan MA, Muller MK, Hahnloser D, Hauri D, Graf R, Clavien PA. The impact of complications on costs of major surgical procedures: a cost analysis of 1200 patients. Ann Surg. 2011 Dec;254(6):907-13. doi: 10.1097/SLA.0b013e31821d4a43. PMID 21562405
- [Background] Spotnitz WD, Burks S. Hemostats, sealants, and adhesives: components of the surgical toolbox. Transfusion. 2008 Jul;48(7):1502-16. doi: 10.1111/j.1537-2995.2008.01703.x. Epub 2008 Apr 14. PMID 18422855
- [Background] Seyednejad H, Imani M, Jamieson T, Seifalian AM. Topical haemostatic agents. Br J Surg. 2008 Oct;95(10):1197-225. doi: 10.1002/bjs.6357. PMID 18763249
- [Background] Sundaram CP, Keenan AC. Evolution of hemostatic agents in surgical practice. Indian J Urol. 2010 Jul;26(3):374-8. doi: 10.4103/0970-1591.70574. PMID 21116358
- [Background] Fok M, Ah-Chong AK, Cheng SW, Wong J. Comparison of a single layer continuous hand-sewn method and circular stapling in 580 oesophageal anastomoses. Br J Surg. 1991 Mar;78(3):342-5. doi: 10.1002/bjs.1800780323. PMID 2021852
- [Background] Scherock TR, Clifford MD, Deveney W, Eneglebert J, Dunphy MD, Factors contributing to leakage of colonic anastomoses, Annual meeting of the Southern Surgical Association Boca Raton, Florida, 1972
- [Background] Lane DA, Philippou H, Huntington JA. Directing thrombin. Blood. 2005 Oct 15;106(8):2605-12. doi: 10.1182/blood-2005-04-1710. Epub 2005 Jun 30. PMID 15994286
- [Background] Tanaka KA, Taketomi T, Szlam F, Calatzis A, Levy JH. Improved clot formation by combined administration of activated factor VII (NovoSeven) and fibrinogen (Haemocomplettan P). Anesth Analg. 2008 Mar;106(3):732-8, table of contents. doi: 10.1213/ane.0b013e318163fc76. PMID 18292410
- [Background] Wheat JC, Wolf JS Jr. Advances in bioadhesives, tissue sealants, and hemostatic agents. Urol Clin North Am. 2009 May;36(2):265-75, x. doi: 10.1016/j.ucl.2009.02.002. PMID 19406326
- [Background] Hung A, Garcia-Tsao G. Acute kidney injury, but not sepsis, is associated with higher procedure-related bleeding in patients with decompensated cirrhosis. Liver Int. 2018 Aug;38(8):1437-1441. doi: 10.1111/liv.13712. Epub 2018 Feb 24. PMID 29393567
- [Background] Randall D, Fenner J, Gillott R, Ten Broek R, Strik C, Spencer P, Bardhan KD. A Novel Diagnostic Aid for Detection of Intra-Abdominal Adhesions to the Anterior Abdominal Wall Using Dynamic Magnetic Resonance Imaging. Gastroenterol Res Pract. 2016;2016:2523768. doi: 10.1155/2016/2523768. Epub 2016 Jan 3. PMID 26880884

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | sFilm-FS | TACHOSIL®
Started | 17 | 16
Completed | 14 | 12
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | sFilm-FS | TACHOSIL® | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.47 (10.46) | 57.81 (19.28) | 60.73 (15.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 9 | 8 | 17
  United States | 3 | 3 | 6
  Slovenia | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus an Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Surgery Through ...
Description: Incidence of Treatment-Emergent Adverse Events AEs related to bleeding at TBS, thrombotic events, transfusion-related complications, post-operative adhesions (MRI assessment)
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population.
Measure: Number; unit: number of TEAEs
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
number of TEAEs
  Total Number of Treatment-Emergent Adverse Events (TEAE) reported | 179 | 168
  Related TEAEs | 0 | 0
  TEAEs leading to discontinuation | 1 | 1
  Serious TEAEs (SAE) | 8 | 6
  Non-fatal serious TEAEs | 7 | 5
  TEAEs leading to death | 1 | 1

2. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Vital Signs
Description: Safety will be assessed from randomization of patients until the last follow-up visit by measuring Systolic Blood Pressure (mmHg)
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
mmHg
  Visit 1 (Screening) from D-21 to D-1 | 137.1 (12.63) | 129.8 (16.75)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 138.9 (11.89) | 133.0 (11.10)
  Visit 3 (Surgery) D0 | 118.9 (20.50) | 111.4 (14.75)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 129.1 (16.97) | 131.4 (21.22)
  Visit 5 (Hospital Discharge) | 133.1 (20.14) | 130.7 (21.08)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 131.6 (13.53) | 123.6 (17.35)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 133.5 (12.52) | 130.0 (15.46)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 130.6 (17.12) | 133.4 (10.34)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 127.0 (19.49) | 134.5 (19.07)

3. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through Physical Examinations
Description: Safety will be assessed from randomization of patients until the last follow-up visit by physical examination: the detection of the number of patients with at least one clinical abnormality in different body areas (abdomen, eyes, skin, cardiovascular)
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Number; unit: number of patients with ≥ 1 abnormality
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
number of patients with ≥ 1 abnormality
  Visit 1 (Screening) from D-21 to D-1 | 6 | 7
  Visit 5 (Hospital Discharge): number analyzed (Participants) | 16 | 16
  Visit 5 (Hospital Discharge) | 3 | 5
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3: number analyzed (Participants) | 15 | 14
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 6 | 5
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3: number analyzed (Participants) | 11 | 7
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 4 | 5
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3: number analyzed (Participants) | 11 | 8
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 6 | 5
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3: number analyzed (Participants) | 16 | 14
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 6 | 4

4. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Urine Analysis Values
Description: Safety will be assessed from randomization of patients until the last follow-up visit by urine analysis (pH)
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
pH
  Visit 1 (Screening) from D-21 to D-1: number analyzed (Participants) | 14 | 15
  Visit 1 (Screening) from D-21 to D-1 | 5.5 (0.60) | 5.9 (0.84)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1): number analyzed (Participants) | 8 | 8
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 5.7 (0.59) | 5.9 (0.88)
  Visit 3 (Surgery) D0: number analyzed (Participants) | 14 | 12
  Visit 3 (Surgery) D0 | 5.4 (0.68) | 5.9 (0.88)
  Visit 5 (Hospital Discharge): number analyzed (Participants) | 11 | 10
  Visit 5 (Hospital Discharge) | 6.2 (1.01) | 6.7 (1.09)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3: number analyzed (Participants) | 13 | 13
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 6.3 (1.01) | 5.8 (0.81)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3: number analyzed (Participants) | 15 | 13
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 5.7 (0.78) | 6.0 (0.90)

5. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Hemoglobin (g/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
g/L
  Visit 1 (Screening) from D-21 to D-1 | 136.1 (20.54) | 135.6 (14.00)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 138.0 (15.13) | 135.0 (15.60)
  Visit 3 (Surgery) D0 | 118.8 (10.64) | 121.9 (12.74)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 104.5 (17.14) | 108.4 (15.96)
  Visit 5 (Hospital Discharge) | 106.8 (16.19) | 111.7 (19.80)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 117.3 (17.02) | 122.1 (15.45)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 118.8 (14.03) | 119.3 (14.66)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 126.8 (12.66) | 128.9 (18.64)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 129.7 (11.66) | 136.3 (18.77)

6. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Detection of Antibodies Against Fibrinogen.
Description: Safety will be assessed from randomization of patients until the last follow-up visit by Measuring plasma levels of antibodies against human fibrinogen, by performing a screening assay using bridging ELISA based on polyclonal antibodies against human fibrinogen, which was developed with a sensitivity of 1000 ng/ml. Patients whose results were above 1000ng/ml control were considered positive.
Time Frame: Last Follow-Up Visit (Visit 9)
Measure: Count of Participants; unit: Participants
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 15 | 13
Participants | 2 | 2

7. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Vital Signs
Description: Safety will be assessed from randomization of patients until the last follow-up visit by measuring Diastolic Blood Pressure (mmHg)
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
mmHg
  Visit 1 (Screening) from D-21 to D-1 | 81.0 (10.59) | 76.0 (7.27)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 75.4 (8.33) | 81.7 (13.61)
  Visit 3 (Surgery) D0 | 61.6 (14.60) | 62.3 (10.87)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 74.2 (12.23) | 75.6 (11.52)
  Visit 5 (Hospital Discharge) | 74.9 (9.50) | 79.9 (11.58)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 79.7 (7.90) | 81.6 (8.45)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 80.8 (9.96) | 81.4 (6.88)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 81.0 (11.86) | 82.7 (7.57)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 79.4 (9.58) | 82.3 (11.56)

8. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Vital Signs
Description: Safety will be assessed from randomization of patients until the last follow-up visit by measuring Heart Rate (beats/minute)
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
beats/minute
  Visit 1 (Screening) from D-21 to D-1 | 72.2 (13.44) | 74.6 (11.94)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 74.5 (12.39) | 79.0 (16.98)
  Visit 3 (Surgery) D0 | 69.0 (19.94) | 79.2 (13.93)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 77.1 (11.17) | 80.9 (18.18)
  Visit 5 (Hospital Discharge) | 79.1 (11.56) | 84.2 (14.87)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 77.3 (16.62) | 78.1 (17.17)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 74.2 (14.26) | 83.1 (8.45)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 73.7 (10.11) | 74.4 (7.61)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 73.7 (16.23) | 73.7 (13.78)

9. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Vital Signs
Description: Safety will be assessed from randomization of patients until the last follow-up visit by measuring Respiratory Rate (breaths/minute)
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
breaths/minute
  Visit 1 (Screening) from D-21 to D-1 | 14.5 (3.14) | 13.5 (1.83)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 14.5 (2.27) | 15.4 (2.56)
  Visit 3 (Surgery) D0 | 15.8 (7.59) | 15.0 (3.13)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 15.0 (2.88) | 16.8 (3.76)
  Visit 5 (Hospital Discharge) | 15.4 (3.12) | 22.4 (27.55)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 13.7 (2.32) | 12.9 (1.00)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 13.1 (1.81) | 14.3 (1.80)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 14.6 (2.29) | 13.4 (1.41)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 13.6 (2.36) | 14.1 (1.44)

10. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Vital Signs
Description: Safety will be assessed from randomization of patients until the last follow-up visit by measuring Body Temperature (°C)
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
°C
  Visit 1 (Screening) from D-21 to D-1 | 36.5 (0.39) | 36.7 (0.33)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 36.6 (0.44) | 36.4 (0.40)
  Visit 3 (Surgery) D0 | 36.4 (0.77) | 36.3 (0.61)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 36.6 (0.44) | 36.8 (0.51)
  Visit 5 (Hospital Discharge) | 36.7 (0.39) | 36.7 (0.52)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 36.4 (0.53) | 36.4 (0.43)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 36.5 (0.34) | 36.8 (0.17)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 36.3 (0.59) | 36.8 (0.20)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 36.5 (0.39) | 36.3 (0.30)

11. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Urine Analysis Values
Description: Safety will be assessed from randomization of patients until the last follow-up visit by urine analysis (Specific Gravity (g/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
g/L
  Visit 1 (Screening) from D-21 to D-1: number analyzed (Participants) | 13 | 12
  Visit 1 (Screening) from D-21 to D-1 | 1021.6 (9.52) | 1018.8 (7.25)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1): number analyzed (Participants) | 8 | 8
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 1017.2 (4.65) | 1019.2 (8.61)
  Visit 3 (Surgery) D0: number analyzed (Participants) | 14 | 12
  Visit 3 (Surgery) D0 | 1027.2 (11.07) | 1022.4 (7.59)
  Visit 5 (Hospital Discharge): number analyzed (Participants) | 11 | 10
  Visit 5 (Hospital Discharge) | 1018.2 (8.94) | 1024.9 (21.39)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3: number analyzed (Participants) | 10 | 9
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 1019.9 (7.62) | 1019.7 (8.96)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3: number analyzed (Participants) | 12 | 8
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 1017.4 (6.02) | 1020.1 (7.61)

12. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Urine Analysis Values
Description: Safety will be assessed from randomization of patients until the last follow-up visit by urine analysis (Presence of Glucose)
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Number; unit: participants
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
participants
  Visit 1 (Screening) from D-21 to D-1 | 6 | 4
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 1 | 0
  Visit 3 (Surgery) D0 | 5 | 4
  Visit 5 (Hospital Discharge) | 7 | 4
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 5 | 4
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 0 | 0
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 0 | 0
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 2 | 3

13. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Mean Cell Hemoglobin Concentration (g/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
g/L
  Visit 1 (Screening) from D-21 to D-1 | 337.3 (15.40) | 337.5 (11.83)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 335.5 (8.14) | 337.5 (8.40)
  Visit 3 (Surgery) D0 | 338.3 (12.16) | 337.7 (12.56)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 336.6 (10.82) | 333.8 (11.41)
  Visit 5 (Hospital Discharge) | 335.9 (10.53) | 333.6 (12.87)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 322.6 (12.02) | 332.1 (12.48)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 324.9 (11.02) | 326.7 (16.71)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 329.8 (11.91) | 326.6 (8.88)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 329.9 (10.77) | 334.9 (15.16)

14. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Mean Cell Hemoglobin (pg))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
pg
  Visit 1 (Screening) from D-21 to D-1 | 29.8 (3.00) | 29.5 (2.27)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 31.3 (2.01) | 28.2 (2.22)
  Visit 3 (Surgery) D0 | 30.4 (1.95) | 29.3 (2.17)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 30.1 (2.11) | 29.6 (2.05)
  Visit 5 (Hospital Discharge) | 30.1 (1.81) | 29.3 (2.45)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 28.7 (2.26) | 29.1 (2.89)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 28.7 (2.38) | 27.5 (3.00)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 28.8 (3.26) | 27.1 (3.10)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 29.4 (2.53) | 29.6 (3.27)

15. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Mean Corpuscular Volume (fL))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
fL
  Visit 1 (Screening) from D-21 to D-1 | 88.5 (6.83) | 87.8 (7.34)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 93.1 (4.70) | 84.3 (8.21)
  Visit 3 (Surgery) D0 | 90.4 (5.84) | 86.8 (6.91)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 89.5 (5.62) | 88.9 (6.35)
  Visit 5 (Hospital Discharge) | 89.9 (4.51) | 87.6 (7.31)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 88.9 (5.43) | 87.9 (8.29)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 88.5 (6.51) | 84.3 (8.79)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 86.9 (7.83) | 82.9 (8.30)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 88.2 (6.96) | 88.8 (9.02)

16. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Red Blood Cell (10^12cells/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: 10^12cells/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
10^12cells/L
  Visit 1 (Screening) from D-21 to D-1 | 4.6 (0.57) | 4.6 (0.53)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 4.4 (0.40) | 4.8 (0.57)
  Visit 3 (Surgery) D0 | 3.9 (0.41) | 4.2 (0.57)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 3.5 (0.58) | 3.7 (0.63)
  Visit 5 (Hospital Discharge) | 3.6 (0.61) | 3.8 (0.66)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 4.1 (0.58) | 4.2 (0.52)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 4.1 (0.43) | 4.4 (0.52)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 4.4 (0.34) | 4.8 (0.63)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 4.5 (0.31) | 4.6 (0.71)

17. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (White Blood Cell (10^9cells/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: 10^9cells/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
10^9cells/L
  Visit 1 (Screening) from D-21 to D-1 | 7.2 (2.47) | 8.0 (2.58)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 8.1 (2.00) | 9.2 (3.21)
  Visit 3 (Surgery) D0 | 11.9 (3.81) | 10.9 (6.43)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 6.43 (4.61) | 12.1 (6.26)
  Visit 5 (Hospital Discharge) | 8.2 (2.93) | 9.6 (5.23)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 6.8 (2.33) | 8.1 (2.01)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 6.2 (3.20) | 7.4 (2.47)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 6.3 (2.56) | 8.0 (2.24)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 8.4 (4.42) | 7.8 (1.53)

18. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Platelet (10^9cells/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: 10^9cells/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
10^9cells/L
  Visit 1 (Screening) from D-21 to D-1 | 241.6 (104.69) | 278.7 (90.90)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 241.6 (82.68) | 308.2 (125.23)
  Visit 3 (Surgery) D0 | 227.4 (100.21) | 275.0 (122.16)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 238.4 (104.66) | 312.6 (173.32)
  Visit 5 (Hospital Discharge) | 308.4 (153.07) | 403.5 (272.79)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 260.9 (111.99) | 330.1 (189.33)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 216.8 (114.38) | 397.3 (204.51)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 203.8 (115.82) | 342.9 (169.86)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 250.2 (98.07) | 276.4 (141.69)

19. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Fibrinogen (g/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
g/L
  Visit 1 (Screening) from D-21 to D-1 | 4.1 (1.16) | 4.3 (1.88)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 3.8 (0.87) | 4.3 (0.82)
  Visit 3 (Surgery) D0 | 3.0 (0.81) | 3.5 (0.63)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 4.9 (1.21) | 5.8 (2.48)
  Visit 5 (Hospital Discharge) | 5.2 (1.10) | 5.8 (2.46)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 4.7 (1.68) | 4.4 (1.88)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 3.7 (0.75) | 4.6 (2.05)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 3.6 (0.95) | 3.6 (0.71)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 3.8 (0.96) | 3.2 (0.47)

20. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (D-Dimer (microg/mL))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: microg/mL
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
microg/mL
  Visit 1 (Screening) from D-21 to D-1 | 1.1 (0.81) | 0.9 (0.90)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 0.8 (0.46) | 1.3 (1.51)
  Visit 3 (Surgery) D0 | 3.8 (3.58) | 2.8 (2.57)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 5.0 (3.32) | 3.3 (1.76)
  Visit 5 (Hospital Discharge) | 4.8 (4.54) | 4.9 (3.69)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 2.3 (1.78) | 2.2 (3.09)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 1.1 (0.68) | 1.3 (1.33)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 1.2 (1.05) | 0.6 (0.30)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 1.4 (2.03) | 4.0 (11.25)

21. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Erythrocyte Sedimentation Rate (mm/hr))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
mm/hr
  Visit 1 (Screening) from D-21 to D-1 | 18.3 (11.60) | 23.7 (18.44)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 20.6 (14.29) | 21.9 (6.85)
  Visit 3 (Surgery) D0 | 17.6 (12.87) | 18.9 (13.30)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 48.5 (25.46) | 53.7 (37.18)
  Visit 5 (Hospital Discharge) | 55.7 (31.99) | 61.9 (41.07)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 39.8 (28.87) | 55.1 (51.17)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 16.5 (10.56) | 46.9 (37.53)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 18.0 (14.13) | 28.1 (18.64)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 17.7 (13.24) | 18.0 (9.86)

22. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (C-Reactive Protein (mg/dL))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
mg/dL
  Visit 1 (Screening) from D-21 to D-1 | 1.1 (1.11) | 1.3 (2.30)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 1.2 (1.46) | 0.9 (0.66)
  Visit 3 (Surgery) D0 | 0.7 (0.90) | 0.7 (0.48)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 8.2 (8.91) | 11.4 (10.02)
  Visit 5 (Hospital Discharge) | 5.6 (5.35) | 5.5 (6.64)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 2.6 (4.97) | 1.6 (2.02)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 0.8 (1.31) | 1.0 (1.17)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 0.5 (0.47) | 0.4 (0.14)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 0.6 (0.86) | 0.5 (0.35)

23. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Blood Urea Nitrogen (mmol/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
mmol/L
  Visit 1 (Screening) from D-21 to D-1 | 5.3 (1.58) | 5.2 (1.28)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 5.8 (1.09) | 4.6 (2.03)
  Visit 3 (Surgery) D0 | 5.1 (1.34) | 4.7 (1.98)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 5.2 (3.98) | 4.9 (2.49)
  Visit 5 (Hospital Discharge) | 4.7 (2.14) | 4.3 (1.73)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 5.1 (2.08) | 4.6 (1.65)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 5.7 (1.53) | 4.1 (1.38)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 5.5 (1.32) | 4.7 (1.55)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 4.2 (1.42) | 4.2 (2.31)

24. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Creatinine (micromol/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
micromol/L
  Visit 1 (Screening) from D-21 to D-1 | 73.6 (18.12) | 61.7 (11.56)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 82.1 (21.02) | 68.9 (10.62)
  Visit 3 (Surgery) D0 | 71.9 (18.48) | 66.5 (19.42)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 67.6 (34.13) | 58.7 (19.73)
  Visit 5 (Hospital Discharge) | 66.7 (19.76) | 59.8 (14.82)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 69.0 (16.50) | 60.0 (7.58)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 71.7 (16.01) | 62.7 (13.46)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 73.4 (21.88) | 65.9 (15.73)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 72.4 (17.81) | 61.6 (9.91)

25. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Uric Acid (micromol/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
micromol/L
  Visit 1 (Screening) from D-21 to D-1 | 434.0 (324.04) | 376.1 (306.72)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 320.4 (84.22) | 346.5 (102.24)
  Visit 3 (Surgery) D0 | 534.2 (585.91) | 401.1 (296.09)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 505.9 (550.82) | 304.8 (153.16)
  Visit 5 (Hospital Discharge) | 426.7 (423.50) | 343.7 (210.83)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 358.1 (307.01) | 431.3 (435.82)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 317.9 (87.80) | 340.0 (59.81)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 321.4 (90.98) | 338.1 (124.09)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 401.6 (345.94) | 312.4 (111.15)

26. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Total Bilirubin (micromol/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
micromol/L
  Visit 1 (Screening) from D-21 to D-1 | 10.9 (6.71) | 12.0 (6.93)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 10.8 (7.62) | 11.6 (4.63)
  Visit 3 (Surgery) D0 | 18.5 (15.69) | 11.6 (6.25)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 16.9 (19.88) | 13.1 (12.01)
  Visit 5 (Hospital Discharge) | 9.8 (6.61) | 8.0 (4.57)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 9.4 (5.11) | 7.1 (2.51)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 8.7 (5.89) | 6.7 (2.15)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 10.1 (5.55) | 7.9 (5.51)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 11.0 (7.60) | 11.3 (6.10)

27. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Lactate Dehydrogenase (microkat/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: microkat/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
microkat/L
  Visit 1 (Screening) from D-21 to D-1 | 3.7 (0.68) | 3.9 (2.28)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 3.6 (0.50) | 3.4 (0.75)
  Visit 3 (Surgery) D0 | 8.1 (6.18) | 5.5 (2.72)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 4.8 (2.30) | 4.6 (1.29)
  Visit 5 (Hospital Discharge) | 4.0 (0.92) | 4.5 (1.19)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 3.5 (0.64) | 3.6 (0.90)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 3.6 (0.44) | 3.7 (1.01)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 3.3 (1.63) | 3.0 (1.60)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 2.9 (0.83) | 3.1 (1.08)

28. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Serum Glutamic Oxaloacetic Transaminase/Aspartate Aminotransferase (microkat/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: microkat/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
microkat/L
  Visit 1 (Screening) from D-21 to D-1 | 0.6 (0.29) | 0.4 (0.23)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 0.5 (0.21) | 0.4 (0.11)
  Visit 3 (Surgery) D0 | 4.2 (4.42) | 1.8 (1.58)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 2.3 (3.42) | 1.2 (1.07)
  Visit 5 (Hospital Discharge) | 0.7 (0.34) | 0.9 (0.62)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 0.5 (0.22) | 0.4 (0.14)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 0.5 (0.30) | 0.5 (0.16)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 0.5 (0.31) | 0.4 (0.24)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 0.5 (0.21) | 0.5 (0.21)

29. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Serum Glutamic Pyruvic Transaminase/Alanine Aminotransferase (microkat/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: microkat/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
microkat/L
  Visit 1 (Screening) from D-21 to D-1 | 0.6 (0.47) | 0.4 (0.23)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 0.4 (0.22) | 0.5 (0.17)
  Visit 3 (Surgery) D0 | 3.2 (3.53) | 1.4 (1.34)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 2.9 (3.86) | 1.4 (1.53)
  Visit 5 (Hospital Discharge) | 0.8 (0.58) | 1.4 (1.28)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 0.7 (1.09) | 0.4 (0.23)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 0.5 (0.41) | 0.4 (0.23)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 0.5 (0.31) | 0.4 (0.14)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 0.5 (0.30) | 0.4 (0.20)

30. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Gamma-GT (microkat/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: microkat/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
microkat/L
  Visit 1 (Screening) from D-21 to D-1 | 2.9 (7.82) | 1.1 (1.10)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 0.6 (0.33) | 0.8 (1.20)
  Visit 3 (Surgery) D0 | 2.8 (7.85) | 0.7 (0.89)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 4.7 (7.43) | 1.1 (0.91)
  Visit 5 (Hospital Discharge) | 3.0 (6.16) | 1.7 (1.23)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 3.8 (7.12) | 1.3 (0.96)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 0.8 (0.82) | 0.8 (0.91)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 0.8 (0.95) | 0.8 (0.85)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 1.2 (1.18) | 0.9 (1.01)

31. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Sodium (mmol/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
mmol/L
  Visit 1 (Screening) from D-21 to D-1 | 141.1 (2.26) | 139.9 (1.89)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 140.0 (3.59) | 139.0 (3.89)
  Visit 3 (Surgery) D0 | 140.9 (2.72) | 139.8 (2.63)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 139.1 (3.19) | 139.7 (2.85)
  Visit 5 (Hospital Discharge) | 139.4 (3.38) | 140.6 (3.07)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 140.9 (2.00) | 139.1 (2.41)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 141.5 (2.54) | 139.9 (2.41)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 140.8 (2.10) | 140.5 (2.78)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 140.3 (1.62) | 140.6 (2.79)

32. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Calcium (mmol/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
mmol/L
  Visit 1 (Screening) from D-21 to D-1 | 2.4 (0.10) | 2.3 (0.16)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 2.4 (0.11) | 2.3 (0.12)
  Visit 3 (Surgery) D0 | 2.1 (0.11) | 2.1 (0.11)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 2.1 (0.14) | 2.1 (0.12)
  Visit 5 (Hospital Discharge) | 2.2 (0.16) | 2.2 (0.13)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 2.5 (0.45) | 3.0 (1.93)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 2.4 (0.11) | 2.4 (0.05)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 2.4 (0.16) | 2.4 (0.10)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 2.4 (0.16) | 2.4 (0.09)

33. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Phosphorous (mmol/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
mmol/L
  Visit 1 (Screening) from D-21 to D-1 | 1.0 (0.12) | 1.1 (0.21)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 1.2 (0.08) | 1.1 (0.16)
  Visit 3 (Surgery) D0 | 1.2 (0.20) | 1.1 (0.33)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 0.9 (0.32) | 0.9 (0.24)
  Visit 5 (Hospital Discharge) | 1.0 (0.19) | 1.0 (0.30)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 1.1 (0.11) | 1.1 (0.19)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 1.1 (0.28) | 1.1 (0.17)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 1.0 (0.24) | 1.1 (0.15)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 1.2 (0.20) | 8.7 (28.57)

34. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Glucose (mmol/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
mmol/L
  Visit 1 (Screening) from D-21 to D-1 | 6.5 (2.51) | 5.6 (1.27)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 6.7 (3.15) | 6.4 (3.78)
  Visit 3 (Surgery) D0 | 8.1 (2.50) | 7.6 (2.65)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 6.1 (1.91) | 6.5 (2.23)
  Visit 5 (Hospital Discharge) | 6.4 (1.62) | 6.0 (1.50)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 6.2 (1.52) | 5.9 (1.91)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 5.9 (1.59) | 6.9 (3.83)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 5.2 (1.73) | 7.1 (5.50)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 6.0 (1.83) | 5.7 (3.37)

35. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Albumin (g/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
g/L
  Visit 1 (Screening) from D-21 to D-1 | 42.4 (4.16) | 42.5 (5.67)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 42.6 (3.89) | 44.0 (4.99)
  Visit 3 (Surgery) D0 | 32.8 (4.77) | 34.5 (4.95)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 28.6 (4.71) | 30.7 (5.08)
  Visit 5 (Hospital Discharge) | 32.4 (5.25) | 34.0 (6.81)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 40.0 (3.35) | 41.1 (4.85)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 41.7 (2.95) | 41.9 (3.93)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 42.9 (4.38) | 44.6 (5.01)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 43.2 (4.71) | 43.8 (4.92)

36. Primary Outcome: To Evaluate the Safety of sFilm-FS Versus the Active-comparator (TACHOSIL®) When Used as Adjunct to Conventional Hemostatic Techniques During Elective Hepatic Surgery Through the Count of Participants With Abnormal Blood / Coagulation Parameters Profiles
Description: Safety will be assessed from randomization of patients until the last follow-up visit by blood/coagulation parameters profiles analysis (Total Protein (g/L))
Time Frame: From visit 1 to visit 9 (an average of 6.5 months)
Population: Descriptive Analysis on Safety Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 17 | 16
g/L
  Visit 1 (Screening) from D-21 to D-1 | 73.2 (5.93) | 73.0 (9.29)
  Visit 2 (Baseline) to be skipped in case Visit 1 is performed one day before surgery (D-1) | 71.1 (5.41) | 74.9 (8.89)
  Visit 3 (Surgery) D0 | 56.6 (8.07) | 62.0 (8.83)
  Visit 4 (Post-Surgery) Daily from D1 to Day of Hospital Discharge | 54.9 (8.68) | 60.5 (10.16)
  Visit 5 (Hospital Discharge) | 63.2 (9.92) | 64.5 (9.60)
  Visit 6 (Follow-up Day 30) D30 (±3) from Visit 3 | 75.0 (6.53) | 76.1 (9.44)
  Visit 7 (Follow-up Day 60) D60 (±7) from Visit 3 | 72.4 (4.99) | 79.3 (8.28)
  Visit 8 (Follow-up Day 120) D120 (±14) from Visit 3 | 75.1 (6.15) | 77.7 (8.10)
  Visit 9 (Follow-up Day 180) D180 (±14) from Visit 3 | 74.8 (6.21) | 75.3 (5.42)

37. Secondary Outcome: To Preliminarily Evaluate the Hemostatic Efficacy of sFilm-FS in Controlling Parenchymal Bleeding During Surgery, Related to Hemostasis and Treatment Failure Through the Proportion of Patients Achieving Hemostasis at TBS
Description: Proportion of patients achieving hemostasis at TBS (absence of bleeding) at 2 (for sFilm-FS product only), 3, 5, 7 or 10 minutes following first product application, without the occurrence of re-bleeding, starting from 10 minutes after product application and until the completion of surgical closure
Time Frame: Day of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 14 | 12
Participants
  2 minutes after application (only for sFilm-FS) | 11 | 0
  3 minutes after application | 12 | 12
  5 minutes after application | 12 | 12
  7 minutes after application | 12 | 12
  10 minutes after application | 14 | 12

38. Secondary Outcome: To Preliminarily Evaluate the Hemostatic Efficacy of sFilm-FS in Controlling Parenchymal Bleeding During Surgery, Related to Hemostasis and Treatment Failure Through the Incidence of Re-treatment at the TBS
Description: Incidence of re-treatment (one or more additional patch of sFilm-FS or TACHOSIL®) at the TBS at the different time points (2 for sFilm-FS, 3, 5, 7, 10 minutes from first product application)
Time Frame: Day of surgery
Population: Descriptive statistics of all randomized patients who underwent surgery, received at least one dose of study treatment and having no major violations of inclusion and exclusion criteria
Measure: Count of Participants; unit: Participants
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 14 | 12
Participants
  2 minutes after application (only for sFilm-FS) | 0 | 0
  3 minutes after application | 0 | 0
  5 minutes after application | 0 | 0
  7 minutes after application | 0 | 0
  10 minutes after application | 2 | 0

39. Secondary Outcome: To Preliminarily Evaluate the Hemostatic Efficacy of sFilm-FS in Controlling Parenchymal Bleeding During Surgery, Related to Hemostasis and Treatment Failure Through the Percentage of Total Patients That Have Achieved Hemostasis
Description: Percentage of total patients (patients that achieved hemostasis with a single patch application and patients that required additional patches) that have achieved hemostasis 10 minutes after first product application and therefore did not need to convert to standard of care treatment at the end of these 10 minutes
Time Frame: Day of surgery
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 14 | 12
Participants | 14 | 12

40. Secondary Outcome: To Preliminarily Evaluate the Hemostatic Efficacy of sFilm-FS in Controlling Parenchymal Bleeding During Surgery, Related to Hemostasis and Treatment Failure Through Incidence of Treatment Failure
Description: Incidence of treatment failure, based on pre-defined treatment failure criteria (in case the bleeding at TBS (or re-bleeding) is still observed after 10 minutes following first application of study product; if hemostasis at TBS is achieved, but the Investigator decides that an additional treatment is required to ensure the durability of hemostasis; if there is a breakthrough bleeding requiring treatment other than the study product, at any time)
Time Frame: Day of surgery
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 14 | 12
Participants | 2 | 0

41. Secondary Outcome: To Preliminarily Evaluate the Hemostatic Efficacy of sFilm-FS in Controlling Parenchymal Bleeding During Surgery, Related to Hemostasis and Treatment Failure.
Description: Incidence of transfusion requirements in the 6 months follow-up period
Time Frame: From surgery, up to 6 months
Population: as for outcome 38
Measure: Number; unit: participants
Arm/Group | sFilm-FS | TACHOSIL®
Number analyzed (Participants) | 14 | 12
participants | 1 | 1

ADVERSE EVENTS:
Time Frame: From Visit 1 to Visit 9 (an average of 6.5 months). All SAE assessed by the Investigator as related to the study drug were continuing to be followed up until 30 days following last visit of the study or until SAE was resolved or stabilized.
Description: Adverse events, especially those related to the study drug were followed up until resolution (returned to baseline status) or stabilization. All AEs were followed-up even after the patient's participation in the study was completed, or in case of withdrawal of the patient from the clinical trial or of anticipated conclusion of the study.
Arm/Group | sFilm-FS | TACHOSIL®
All-Cause Mortality (participants affected / at risk) | 1/17 | 1/16
Serious Adverse Events (participants affected / at risk) | 6/17 | 5/16
Other Adverse Events (participants affected / at risk) | 17/17 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | sFilm-FS (N=17) | TACHOSIL® (N=16)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 1 (1)
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 2 (2) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
DISEASE PROGRESSION (General disorders) | 1 (1) | 0 (0)
IMPAIRED HEALING (General disorders) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
MALNUTRITON (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MUSCLE AROPHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | sFilm-FS (N=17) | TACHOSIL® (N=16)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
BLOOD LOSS ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
COAGULOPATHY (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
IRON DEFICIENTY ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (3) | 1 (2)
ATRIAL TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
COR PULMONALE (Cardiac disorders) | 0 (0) | 1 (1)
CARDIOMEGALY (Cardiac disorders) | 1 (1) | 0 (0)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 1 (1)
PERICARDIAL CYST (Cardiac disorders) | 1 (1) | 0 (0)
RIGHT VENTRICULAR ENLARGEMENT (Cardiac disorders) | 0 (0) | 1 (1)
RIGHT VENTRICULA FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 2 (2) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
SYSTOLIC DYSFUNCTION (Cardiac disorders) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 1 (2) | 3 (4)
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICULA EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICULAR HYPOKINESIA (Cardiac disorders) | 0 (0) | 1 (1)
FACTOR II DEFICIENCY (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 2 (3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (3) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 0 (0)
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 2 (2) | 2 (2)
ABNORMAL FAECES (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 3 (3) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 2 (5)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
DUODENITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
INFLAMMATORY BOWEL DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTRA ABDOMINAL HAEMATOMA (Gastrointestinal disorders) | 1 (1) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 12 (14) | 5 (5)
VOMITING (Gastrointestinal disorders) | 2 (2) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 1 (2)
CHEST PAIN (General disorders) | 1 (1) | 1 (1)
DEATH (General disorders) | 0 (0) | 1 (1)
DISEASE PROGRESSION (General disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0)
GENERALISED OEDEMA (General disorders) | 0 (0) | 1 (2)
IMPAIRED HEALING (General disorders) | 1 (1) | 1 (1)
INFLAMMATORY PAIN (General disorders) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 2 (5)
PAIN (General disorders) | 3 (4) | 5 (11)
PYREXIA (General disorders) | 2 (2) | 3 (3)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATORENAL FAILURE (Hepatobiliary disorders) | 1 (1) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (2) | 0 (0)
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 0 (0) | 1 (1)
ABDOMINAL INFECTION (Infections and infestations) | 2 (2) | 0 (0)
BACTERIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CANDIDA INFECTION (Infections and infestations) | 1 (1) | 1 (1)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
INFECTION SUSCEPTIBILITY INCREASED (Infections and infestations) | 1 (2) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1)
POST PROCEDURAL INFECTION (Infections and infestations) | 1 (2) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 2 (3) | 3 (5)
CONFUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
DRAIN SITE COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEPATIC SEROMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LUMBAR VERTEBRAL BILE LEAK (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL BILE LEAK (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 11 (13) | 9 (11)
SEROMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD ALBUMIN INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD BILIRUBIN INCREASE (Investigations) | 1 (1) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 (1) | 0 (0)
GAMMA GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 (2) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
FOLATE DEFICIENCY (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 8 (12) | 5 (5)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOPHAGIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
MAGNESIUM DEFICIENCY (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCLE ATRHOPHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
ADRENAL GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CHOLANGIOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
GALLBLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
HAEMANGIOMA OF SPLEEN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NEUROENDOCRINE CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COGNITIVE DISORDER (Nervous system disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 2 (2)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 2 (2)
LETHARGY (Nervous system disorders) | 0 (0) | 1 (1)
POLYNEUROPATHY (Nervous system disorders) | 1 (2) | 0 (0)
RADICULOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
AGITATION (Psychiatric disorders) | 2 (2) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 1 (1)
INSOMNIA (Psychiatric disorders) | 2 (2) | 1 (1)
RESTLESSNESS (Psychiatric disorders) | 1 (1) | 1 (1)
SLEEP DISORDER (Psychiatric disorders) | 3 (3) | 2 (3)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2) | 3 (3)
OLIGURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL INFARCT (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1)
GENITAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PENILE HAEMATOMA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PENILE PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
EXCESSIVE GRANULATION TISSUE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
LIPODYSTROPHY ACQUIRED (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
PRURITUS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
BLOOD VOLUME EXPANSION (Surgical and medical procedures) | 0 (0) | 1 (1)
COLONIC LAVAGE (Surgical and medical procedures) | 1 (1) | 0 (0)
DERMABRASION (Surgical and medical procedures) | 0 (0) | 1 (1)
HAEMATOMA EVACUATION (Surgical and medical procedures) | 1 (1) | 0 (0)
PROPHYLAXIS (Surgical and medical procedures) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 3 (3) | 2 (2)
HYPOTENSION (Vascular disorders) | 2 (3) | 2 (5)
INFERIOR VENA CAVA DILATATION (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT04660721/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT04660721/SAP_001.pdf